CLINICAL TRIAL: NCT07272161
Title: Pilot Evaluation of the StarGuide Next Generation SPECT/CT System
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Carrie Hruska, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 25-010203
Record Dates: First submitted 2025-11-24; First posted 2025-12-09 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-02

CONDITIONS: Nuclear Medicine
Keywords: SPECT/CT

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Nuclear medicine imaging (Experimental): Participants presenting to Nuclear Medicine for clinically-indicated administration of radiopharmaceuticals and imaging tests on approved clinical scanners will undergo an additional scan for research purposes on the investigational StarGuide NextGen system.
  Interventions: Device: StarGuide NextGen SPECT/CT system

INTERVENTIONS:
Device: StarGuide NextGen SPECT/CT system — Within 1 hour of the participant receiving a scheduled clinical nuclear medicine procedure, a research scan will be performed with the StarGuide NextGen SPECT/CT system for detection of radiopharmaceutical uptake in the patient body. The total time for the scan will range from 20 - 60 minutes.

SUMMARY:
The goal of this pilot study is to evaluate capabilities of the StarGuide NextGen SPECT/CT system to inform future clinical use of this technology.

DETAILED DESCRIPTION:
The StarGuide NextGen system is expected to offer superior image quality and faster scanning times relative to our standard clinical SPECT systems. However, the optimal scanning parameters for StarGuide NextGen are yet undetermined. This research study is necessary to assess the feasibility of patient scanning on this system and to refine the parameters in preparation for future clinical use. The study is also important to inform whether and to what degree the StarGuide NextGen can improve image quality over standard dual-head SPECT/CT scanners for a variety of common nuclear medicine exams.

ELIGIBILITY:
Inclusion Criteria:

* Scheduled for clinical administration of a radiopharmaceutical for a clinical nuclear medicine imaging test or radiopharmaceutical therapy
* Able to provide consent for study participation StarGuide NextGen Evaluation

Exclusion Criteria:

* Unable to comply with physical requirements for lying supine on the StarGuide NextGen patient bed
* Pregnant. (Note that pregnancy status will be established via clinical standard of care for the clinical nuclear medicine test prior to administration of radiopharmaceutical.)
* Unable to provide consent for study participation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2027-01 (Estimated); Study Completion 2027-01 (Estimated)

PRIMARY OUTCOMES:
Diagnostic image quality | 1 year
  Diagnostic image quality of StarGuide NextGen and clinical scans, will be assessed by study radiologists using a Likert scale of 1-5, where 1 = Non-diagnostic; 2 = Poor; 3 = Adequate; 4 = Good; and 5 = Excellent. For future clinical use, acceptable image quality will be considered as having scores of 4 or 5.

SECONDARY OUTCOMES:
Count sensitivity | 1 year
Lesion contrast | 1 year
Signal-to-noise ratio (SNR) | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Carrie B. Hruska, PhD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No